CLINICAL TRIAL: NCT02119208
Title: Effects of the Intensity and the Timing of the Physical Activity in a Primary School
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Marie-Ève Mathieu, Assistant professor, Université de Montréal
Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-135-CERES-P
Record Dates: First submitted 2014-02-23; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Energy Intake

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: Intensity and timing of exercise

INTERVENTIONS:
Behavioral: Intensity and timing of exercise

SUMMARY:
1. In natural environment, the moderate-intensity break will allow a reduction of the caloric intake at the dinner more important than for the light-intensity break
2. In natural environment, the break taken juste before dinner will allow a reduction of the caloric intake at the diner more important than earlier in the day.

ELIGIBILITY:
Inclusion Criteria:

* Children aged of approximately 5 years old of a of a nursery class of the school Jacques-Barclay, St-Mathieu

Exclusion Criteria:

* Present allergy of the foods in the lunch
* having a handicap or a limitation that avoid walking, running or tkaing part of the physcial activity courses at the school.
* Having a potential surgery
* Having a metabolic disease or taking drugs that could have an impact on the results of the study
* Be vegetarian
* Having intestinal disorders

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Caloric intake at the breakfast, lunch and diner (kj) | 3 days per condition

SECONDARY OUTCOMES:
Anthropometric measures | At preliminary visit

CONTACTS AND LOCATIONS:
Locations (1):
- École Jacques-Barclay, Saint-Mathieu, Quebec, Canada